CLINICAL TRIAL: NCT07042646
Title: The Effect of Sexual and Reproductive Health Training on Sexual Function and Quality of Sexual Life in Women With Physical Disabilities: A Pilot RCT Study From a Turkiye Perspective
Brief Title: Sexual Function and Quality of Sexual Life in Women With Physical Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Gozde Yıldız Daş Geçim, Assist. Prof., Amasya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Amasya32
Record Dates: First submitted 2025-06-18; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Disability Physical
Keywords: women with physically disabled; sexual health; psychosexual dysfunctions; sexuality
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Sexuality | interventions — Sex

STUDY DESIGN:
Intervention Model Description: a randomised controlled trial : a pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Sexual and Reproductive Health Training program received the intervention group.
  Interventions: Behavioral: Sexual and Reproductive Health Training program
- Control group (No Intervention): no intervention was the control group.

INTERVENTIONS:
Behavioral: Sexual and Reproductive Health Training program — 'The Sexual and Reproductive Health education program was prepared by researchers who are experts in the field of public health and public health nursing. The program was implemented once a week for 3 weeks (why 3 weeks) in 50-60 minute sessions (Table 1). The content and duration of the application were prepared in accordance with the Ministry of Health Sexual and Reproductive Health: National Strategic Action Plan for the Health Sector (2005-2015) and the Turkey Reproductive Health Program Sexual and Reproductive Health Service Standards (2007). Each program session was two education sessions, and all the questions of the disabled woman were answered .
  Arms: Intervention group

SUMMARY:
This pilot randomized controlled trial will be carried out with women with physical disabilities registered at a disability center. A total of 49 participants will be randomly assigned to either the intervention group or the control group. Following a three-week follow-up period, the study will be completed, with a total of 26 participants: 16 in the intervention group and 10 in the control group . SRH training will be provided to the intervention group once a week, for a total of three sessions. At the beginning and end of the study, both groups will be administered a survey including demographic information, the Sexual Quality of Life Questionnaire-Female (SQLQ-F), and the Female Sexual Function Index (FSFI).

DETAILED DESCRIPTION:
Background: Ensuring that women with disabilities, who are among disadvantaged groups, maintain and improve their sexual and reproductive health (SRH) on equal terms with other women is of great importance. The purpose of this study is to examine the impact of SRH training provided to women with physical disabilities on their sexual function and quality of sexual life, as well as to assess the feasibility and acceptability of the educational intervention.

Method: This pilot randomized controlled trial will be carried out with women with physical disabilities registered at a disability center. A total of 49 participants will be randomly assigned to either the intervention group or the control group. Following a three-week follow-up period, the study will be completed, with a total of 26 participants: 16 in the intervention group and 10 in the control group . SRH training will be provided to the intervention group once a week, for a total of three sessions. At the beginning and end of the study, both groups will be administered a survey including demographic information, the Sexual Quality of Life Questionnaire-Female (SQLQ-F), and the Female Sexual Function Index (FSFI).

ELIGIBILITY:
Inclusion Criteria:

* Those who were female between the ages of 18-65, physically disabled, married, did not have a mental health problem, did not have a communication barrier, and volunteered were included in this study.

Exclusion Criteria:

* being a man
* having a disability other than physical disability

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2024-09-14 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Quality of Sexual Life | 1 months
  The scale has 6 sub-dimensions: desire, arousal, lubrication, orgasm, satisfaction, and pain (Rosen et al., 2000). Each item is scored from 0 to 5. The highest score that can be obtained from the scale is 95.0, and the lowest score is 4.0.

SECONDARY OUTCOMES:
Sexual Function | 1 months
  The scale is suitable for women aged 18 and over, is a six-point Likert type, and consists of 18 items. Each item is answered by considering the sexual life in the last four weeks. The original version of the scale states that each item can be scored between 1-6 or 0-5. In this study, a 1-6 point system was used (1=I completely agree, 2=I largely agree, 3=I partially agree, 4=I partially disagree, 5=I largely disagree, 6=I completely disagree). The highest score that can be obtained from the scale in the 1-6 point system is 108, and the lowest score is 18.

CONTACTS AND LOCATIONS:
Overall Officials: zehra incedal sonkaya, PhD, Study Chair — Amasya University; murat yücel, PhD, Study Chair — Amasya University
Locations (1):
- Amasya University Faculty of Health Sciences, Amasya, Turkey (Türkiye)